CLINICAL TRIAL: NCT05522712
Title: Acapella Versus Incentive Spirometer on Cardiopulmonary Fitness After Heart Valve Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samira Abdelrehim Mahmoud shehata, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003310
Record Dates: First submitted 2022-08-20; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Open Heart Surgery; Heart Valve Diseases; Heart Diseases
MeSH Terms: conditions — Heart Valve Diseases; Heart Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acapella user (Experimental): this group will use acapella in addition to traditional chest physiotherapy , early mobility and sternal precautions.
  Interventions: Device: Acapella user
- Incentive spirometer user (Experimental): this group will receive incentive spirometer in addition to traditional chest physiotherapy, early mobility and sternal precautions.
  Interventions: Device: Incentive spirometer user
- Control user (Other): this group will receive traditional chest physiotherapy , early mobility and sternal precautions.
  Interventions: Procedure: Control

INTERVENTIONS:
Device: Acapella user — The exercise session will include three sets of deep breaths. Each set will include 10 repetitions which were fol¬lowed by 30 to 60 seconds pause in between. Patients will be instructed to perform slow maximal inspiration, while expiration was done through acapella in a prolonged manner to minimize airway closure and alveolar collapse. In the Acapella device, resistance was increased continuously on each successive day. The technique will be applied for 15 minutes.
  Components of Acapella® treatment will include :
  * Breathing control
  * 10 breaths through the Acapella® device
  * Inhaling up to approximately three - quarter maximum breathing capacity
  * 2-3 second breath hold
  * Active exhalation to Functional residual capacity but not too forcefully (3-4 second)
  * The patient did 2-3 huffs at the end of the session, Cough or forced expiration in a set cycle.
  Arms: Acapella user
Device: Incentive spirometer user — 1. Sit upright in a chair or in bed. Hold the incentive spirometer at eye level, hold a pillow to help splint or brace the incision to decrease pain at incision.
  2. Put the mouthpiece in mouth and close lips tightly around it. Slowly breathe out (exhale) completely.
  3. Breathe in (inhale) slowly through mouth as deeply as possible. As taking the breath, the ball will rise.
  4. Try to get the ball as high as possible.
  5. When getting it, hold breath for 10 seconds, or as long as possible.
  6. Then, breathe out slowly through mouth. Then, Rest for a 30-60 seconds.
  7. Repeat 10 times. Try to get the ball to the same level or higher with each breath.
  8. repeat 10 times for 3 sets.
  Arms: Incentive spirometer user
Procedure: Control — This group is a control group will not receive new intervention just traditional chest physiotherapy and mobilization
  Arms: Control user

SUMMARY:
Valvular heart disease (VHD) is a growing and important public health problem due to the increasing prevalence of degenerative VHD, accompanied by prolonged life expectancy in developed countries. It is associated with high morbidity and mortality.Heart valve surgery is one of the proven treatments of VHD, which corrects hemodynamic abnormalities that could contribute to decrease mortality and improvement in quality of life, despite the improvement in the hemodynamic parameters, the cardiorespiratory fitness level remained low after heart valve surgery.

Cardiac surgeries can cause a series of clinical and functional complication. Postoperative pulmonary complications are the most common, in turn, contribute directly to increase morbidity and mortality and longer hospital stays.Mucociliary clearance is affected after open-heart surgery by the effects of general anaesthesia, intubation and analgesia. Expiratory flow rate is directly related to lung volume and therefore when lung volumes are decreased, coughing will be less effective.

Chest physical therapy plays an important role in the prevention and management of postoperative pulmonary complications. It includes deep breathing exercises, mobilization, postural drainage, percussion and vibration or shaking which were developed to improve bronchial drainage. Airway clearance techniques are commonly used for clearing secretions, improving gas exchange, oxygenation, and work of breathing. Acapella® is an airway clearance device that combines the resistive features of a positive expiratory pressure device with oscillations which diminishes the mucus adhesiveness and decrease the collapsibility of airways.

In the present study, the aim is to compare the effect of acapella and incentive spirometer on cardiopulmonary fitness in patients undergoing heart valve surgery. Those patients may gain a more benefit from acapella application and incentive spirometer so, prevent post-operative pulmonary complication, reduce hospitalization and hospital costs, and improve quality of life. Therefore, early mobilization and chest physiotherapy including acapella and incentive will be started on 1st day after discharge from cardiac care unit (CCU) .

DETAILED DESCRIPTION:
This study is designed to compare between effect of acapella and incentive spirometer on cardiopulmonary fitness after heart valve surgery.The patients of this study will randomly assigned into three equal groups in numbers.

Study Group A will receive acapella protocol in addition to traditional chest physiotherapy, early mobilization and sternal precautions.

Study Group B will receive incentive spirometer in addition to traditional chest physiotherapy, early mobilization and sternal precautions.

Control Group C will receive traditional chest physiotherapy, early mobilization and sternal precautions.

The program of treatment for each patient will be applied daily starting from the first day the patient will be extubated (2nd postoperative day) up to 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with age ranges (30-40) years old.
* Patients with normal body mass index ranges (18.5-24.9) kg/m2
* Patients undergo mitral valve surgery via median sternotomy.
* Post operative, extubated heart valve surgery patients, who were able to follow the instructions and sign the consent form.
* Patients with hemodynamic stability.
* Patients with controlled diabetes mellitus.

Exclusion Criteria:

* - Patients who required more than 48 hours of intubation after surgery.
* Reintubation in post operative period.
* Patients who had history of respiratory tract infection within a period of three months.
* Patients undergo CABG ,or double valve surgery.
* Patients with any neuromuscular disease.
* Patients with severe renal dysfunction.
* Anemic patients.
* Uncontrolled diabetes mellitus.

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function test | 7 days
  Forced vital capacity and forced expiratory volume in one second will be measured
Peripheral oxygen saturation | 7 days
  Determine level of oxygen in blood
Rate of perceived exertion | 7 days
  Dysnpea level measured by modified borg scale from 0 to 10 0 no dyspnea at all 10 maximal degree of dyspnea
Pain intensity | 7 days
  Measured by visual analogue scale to determine degree of incisional pain 0 no pain 10 worst pain
Cardiorespiratory fitness evaluation | 7 days
  Vo2max is measured to determine functional capacity after operation
Length of hospital stay | Average 4 - 7 days
  Determine how many days patient need to be in hospital and become fully hemodynamically stable

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab M. Helmy, PhD, Study Chair — Cairo University
Locations (1):
- Faculty of physical therapy, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No